CLINICAL TRIAL: NCT06510049
Title: Validity and Reliability of Ultrasound Imaging for Measuring Coronal and Sagittal Angles in Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KS-467-01
Record Dates: First submitted 2024-06-30; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Ultrasonography; Coronal; Sagittal; Idiopathic Scoliosis; Validation Studies as Topic; Program Evaluation
Keywords: Ultrasonography; Coronal; Sagittal; Idiopathic Scoliosis; Reliability; Validity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with idiopathic scoliosis (IS), especially children and adolescents, require regular follow-up evaluations. Ultrasound imaging offers a reliable, radiation-free method for assessing spinal curvatures in the coronal and sagittal planes. While manual labeling in traditional ultrasound is error-prone, automated labeling reduces inaccuracies but still needs further validation, particularly in the sagittal plane. This study compared three-dimensional (3D) ultrasound assessments with conventional X-ray images--the clinical gold standard. And it is aimed to evaluate the validity and reliability of ultrasound measurements-Ultrasound Curve Angle (UCA) and Ultrasound Lamellar Angle (USLA)-against established radiographic benchmarks like Cobb's angle, Thoracic Kyphosis (TK), and Lumbar Lordosis (LL).

DETAILED DESCRIPTION:
This study was structured into two fundamental segments: 1) a dual-operator analysis focused on evaluating both intra- and inter-operator reliability of the UCA and USLA; and 2) a validation study of radiographic indices, specifically the coronal Cobb angle, TK, and LL, in correlation with UCA and USLA measurements. Initially, 100 patients diagnosed with IS were subjected to both standard radiographic and 3D ultrasound examinations. Owing to various exclusion criteria, 20 patients were subsequently disqualified from the study, resulting in a final sample of 80 patients for statistical evaluation. Reliability assessments were conducted using the Intraclass Correlation Coefficient (ICC). Furthermore, the validity of the UCA and USLA measurements was rigorously analyzed by comparing them against established radiographic benchmarks, utilizing Pearson correlation coefficients and Bland-Altman plots for comprehensive evaluation. All expected or unexpected adverse events from this study will be recorded and monitored.For comprehensive analysis, participants were systematically categorized based on multiple demographic and clinical parameters: coronal angle (either ≥20° or <20°), gender (male or female), age (either>14 years or ≤14 years), and nutritional status (classified as normal or abnormal).

ELIGIBILITY:
Inclusion Criteria:

* Patients with IS who were cooperative with ultrasound procedures.

Exclusion Criteria:

* Patients with spinal disorders such as Marfan's syndrome, a history of ankylosing spondylitis, or spinal neurofibroma.
* Patients with severe medical or psychiatric conditions that could potentially impact the study results.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with IS who have been admitted to the Scoliosis Traditional Chinese and Western Medicine Diagnosis and Treatment Center of Zhejiang Provincial Hospital of Traditional Chinese Medicine since May 2023.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Coronal thorax/thoracolumbar/lumbar cobb angle and sagittal thorax/thoracomaxillary/lumbar anterior and posterior lordosis angles on x-ray | January to May 2024
  Coronal thorax/thoracolumbar/lumbar cobb angle and sagittal thorax/thoracomaxillary/lumbar anterior and posterior lordosis angles on x-ray
Coronal thoracic/thoracolumbar/lumbar cobb angle and sagittal thoracic/thoracomaxillary/lumbar anterior-posterior lordosis angle on ultrasound | January to May 2024
  Coronal thoracic/thoracolumbar/lumbar cobb angle and sagittal thoracic/thoracomaxillary/lumbar anterior-posterior lordosis angle on ultrasound

SECONDARY OUTCOMES:
gender | January to May 2024
  gender
age | January to May 2024
  age
BMI | January to May 2024
  BMI

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine (Zhejiang Provincial Hospital of Traditional Chinese Medicine), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No